CLINICAL TRIAL: NCT00448032
Title: A Multiple Ascending Dose Study of the Safety, Tolerability, and Pharmacokinetics of Ppm-204 Administered Orally to Healthy Male Japanese Subjects
Brief Title: Study Evaluating Multiple Oral Doses of PPM-204 in Healthy Japanese Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: 3180A1-107
Record Dates: First submitted 2007-03-14; First posted 2007-03-15 (Estimated); Last update posted 2007-12-05 (Estimated); Status verified 2007-12

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

INTERVENTIONS:
Drug: PPM-204

SUMMARY:
A study evaluating the safety and pharmacokinetics of multiple oral doses of an investigational oral diabetic agent when given to healthy Japanese male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Men, aged 20 to 45 years, inclusive
* Body mass index in the range of 17.6 to 26.4 kg/m2
* Healthy as determined by the investigator on the basis of medical history, physical examination, clinical laboratory test results, vital signs, and 12-lead electrocardiogram (ECG)

Exclusion Criteria:

* History of cardiac, thyroid, muscle, and kidney abnormalities
* History of NSAID induced bronchospasm or asthma
* History of any clinically important allergies

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2006-11; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Safety

SECONDARY OUTCOMES:
Pharmacokinetics/Pharmacodynamics

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Tokyo, Japan